CLINICAL TRIAL: NCT02836665
Title: Application of Telemedicine for Dermatological Emergency Patients
Acronym: Telederm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-033
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dermatological Emergency
Keywords: Emergency Room; Manchester Triage System; Telemedicine; Patients
MeSH Terms: conditions — Emergencies | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Control group (No Intervention): Patients of group A wait routinely until the dermatological investigator in charge arrives at the emergency room. Once the dermatological investigator is on site, he gives a diagnosis and proposes a therapy.
- B: Telemedicine for dermatological emergency patients (Experimental): For Patients of group B study-related photographs of the skin lesion and anamnesis data are uploaded to the hospital information system "medico". Those data can directly be processed by the dermatological investigator in charge who enters his diagnosis and his therapy proposal.
  Interventions: Procedure: Telemedicine for dermatological emergency patients

INTERVENTIONS:
Procedure: Telemedicine for dermatological emergency patients — Study-related photographs of the skin lesion made by a tablet and anamnesis data are uploaded to the hospital information system "medico". Those data can directly be processed by the dermatological investigator in charge who enters his diagnosis and his therapy proposal without being on site.
  Arms: B: Telemedicine for dermatological emergency patients

SUMMARY:
After admission to the emergency room each dermatological patient is routinely assessed to Manchester Triage System (MTS) by the nursing staff. Thereby data are collected for anamnesis followed by randomization in two equal study groups.

Patients of group A (control group) wait routinely until the dermatological investigator in charge arrives at the emergency room. Once the dermatological investigator is on site, he gives a diagnosis and proposes a therapy.

For Patients of group B (teledermatology) study-related photographs of the skin lesion and anamnesis data are uploaded to the hospital information system "medico". Those data can directly be processed by the dermatological investigator in charge who enters his diagnosis and his therapy proposal.

Subsequently an internal control is carried out as the same investigator comes personally to the emergency room to check its telemedical diagnosis and therapy proposal.

Finally both time periods patients have to wait in the emergency room for their diagnosis and therapy are compared with each other.

DETAILED DESCRIPTION:
After admission to the emergency room each dermatological patient is routinely assessed to Manchester Triage System (MTS) by the nursing staff. Thereby data are collected for anamnesis (duration of symptoms, allergies, self-medication, medical history) followed by randomization in two equal study groups.

Patients of group A (control group) wait routinely until the dermatological investigator in charge arrives at the emergency room. Once the dermatological investigator is on site, he gives a diagnosis and proposes a therapy.

Time is measured from the patients admission to the emergency room up to the personnel diagnosis and therapy by the dermatological investigator in charge.

For Patients of group B (teledermatology) first of all study-related photographs of the skin lesions are taken with a tablet. After that the registration of the consult "teledermatology" is carried out by the emergency investigator in charge, who uploads the photographs as well as the data for anamnesis to the hospital information system "medico". The consult "teledermatology" can directly be processed by the dermatological investigator in charge who enters his diagnosis and his therapy proposal.

Time is measured from admission to the emergency room up to the telemedical diagnosis and therapy by the dermatological investigator in charge.

Subsequently an internal control is carried out as the same investigator comes personally to the emergency room to check its telemedical diagnosis and therapy proposal.

Finally both time measurements are compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Written informed consent prior to study participation
* Adults who are contractually capable and mentally able to understand and follow the instructions of the study personnel.
* Dermatological emergency patient

Exclusion Criteria:

* Male or female aged < 18 years
* Missing informed consent prior to study participation
* Patient has been committed to an institution by legal or regulatory order
* Persons in dependence from the sponsor or working with the sponsor
* Participation in another clinical trial within the previous 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Waiting time [min] | 1 emergency visit [approximately 2 hours]
  Time is measured from the patients admission to the emergency room up to the personnel/telemedical diagnosis and therapy by the dermatological investigator in charge.

SECONDARY OUTCOMES:
Number of differences between the personally and the telemedical diagnosis and therapy proposal | 1 emergency visit [approximately 2 hours]
  An internal control is carried out as the same investigator comes personally to the emergency room to check its telemedical diagnosis and therapy proposal.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Villa, Dr. med., Principal Investigator — RWTH Aachen University
Locations (1):
- Uniklinik RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marsden J, Windle J, Mackway-Jones K. Emergency triage. Emerg Nurse. 2013 Jul;21(4):11. doi: 10.7748/en2013.07.21.4.11.s11. No abstract available. PMID 23901863